CLINICAL TRIAL: NCT05701683
Title: IMPROVEMENT in ERADICATION of H-PYLORI INFECTION With ADDITION of LACTOBACILLUS REUTERI
Brief Title: IMPROVEMENT in ERADICATION of H-PYLORI INFECTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Dr.Mehreen Akmal, Principal Investigator, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0493-2019-LNH-ERC
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Lactobacillus reuteri; Helicobacter pylori; Dyspepsia; Eradication Therapy
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ERADICATION of H-PYLORI INFECTION with ADDITION of LACTOBACILLUS REUTERI (Experimental): In experimental group, patients receiving clarithromycin based sequential therapy with LACTOBACILLUS REUTERI
  Interventions: Drug: Lactobacillus Reuteri Probiotic
- ERADICATION of H-PYLORI INFECTION without LACTOBACILLUS REUTERI (No Intervention): control group included patients who received clarithromycin based sequential therapy alone

INTERVENTIONS:
Drug: Lactobacillus Reuteri Probiotic — Experimental group receiving Lactobacillus Reuteri Probiotic with sequential therapy
  Other Names: sequential therapy with Lactobacillus Reuteri Probiotic
  Arms: ERADICATION of H-PYLORI INFECTION with ADDITION of LACTOBACILLUS REUTERI

SUMMARY:
Efficacy in terms of H pylori eradication of clarithromycin based sequential therapy with lactobacillus is better than sequential based therapy alone.

DETAILED DESCRIPTION:
Data Collection:

Subjects attending outpatient in department of Gastroenterology meeting the inclusion & exclusion criteria in Liaquat National Hospital, Karachi with H. pylori related chronic gastritis with/without peptic ulcers on endoscopy & gastric biopsy (histopathology) or Stool for H. pylori antigen +ve, or Rapid urease test +ve or Positive Urea Breath Test as per operational definition will be included. For all patients included in this study, we will collect the following information age, gender, duration of the disease.Patients will be divided into two groups randomly, group A and B.In group A (case) patients along with standard sequential therapy :

* Amoxil 1000 mg twice daily for first 5 days
* clarithromycin 500 mg twice daily plus Tinidazole 500 mg twice daily for next 5 days with addition of lactobacillus R 100 mg twice daily in capsule form will be given for 2 weeks. While group B (control) will include patients who have already received standard sequential therapy which is
* Amoxil 1000mg twice daily for first 5 days
* Clarithromycin 500 mg twice daily plus Tinidazole 500 mg twice daily for next 5 days After completion of 6 weeks of proton pump inhibitors (PPI), it will be stopped. As per our protocol for all patients , after 1-2 weeks of stopping PPI stool sample will be collected and will be sent to the laboratory of the institute for helicobacter pylori stool antigen (HPSA).This test is performed as routine to check the success of eradication therapy. H. pylori eradication will be achieved if post treatment HPSA is negative. All demography, clinical history will be recorded by a principal investigator on a predesigned proforma, informed written consent will be taken before enrolment. Exclusion criteria will be followed strictly to avoid confounding variables.

MATERIAL AND METHODS

Study design:

Randomized control study.

Setting:

Study was conducted in Out Patients Department of Gastroenterology, Liaquat National Hospital, Karachi.

Duration: One year after approval of synopsis from hospital ethics committee.

Sample size:

Sample size: Sample size was calculated on the basis of the following eradication rate of H. Pylori with clarithromycin based sequential therapy regimen was= 76%(no relevant statistics available regarding combination of clarithromycin based sequential therapy regimen with lactobacillus Reuteri) Confidence level=95% Bond on error= 6% Sample size (n) = 195 no: of H. Pylori positive Patients in each group, with total of 390 patients Formula n= z2p (1-P) /d2

Inclusion criteria:

* Patients between 18 years to 60 years of age.
* Either gender
* Patients having H. pylori related chronic gastritis with/without peptic ulcers on endoscopy & gastric biopsy (histopathology) or Stool for H. pylori antigen +ve , or Rapid urease test +ve

Exclusion criteria:

* Pregnant women
* End stage renal disease (GFR <15 mL/min/)
* Chronic Liver Disease

Data analysis:

Statistical package for Social Sciences (SPSS version 22) was used for data analysis. Frequencies and percentages were computed for qualitative variables like gender, post eradication HPSA (negative/positive). Quantitative variables will be presented as mean ± standard deviation for age and duration of dyspepsia. Effect modifiers like age, gender, duration of dyspepsia were controlled through stratification. Post stratification Chi-square test was used. P value ≤0.05 was considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 years to 60 years of age.
* Either gender
* Patients having H. pylori related chronic gastritis with/without peptic ulcers on endoscopy & gastric biopsy (histopathology) or Stool for H. pylori antigen +ve , or Rapid urease test +ve

Exclusion Criteria:

* Pregnant women
* End stage renal disease (GFR <15 mL/min/)
* Chronic Liver Disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Eradication rate | 8 weeks after therapy
  eradication of helicobacter pylori infection after 8 weeks of completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mehreen Akmal, MBBS, Principal Investigator — Liaquat National Hospital & Medical College
Locations (1):
- Mehreen Akmal, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eslami M, Yousefi B, Kokhaei P, Jazayeri Moghadas A, Sadighi Moghadam B, Arabkari V, Niazi Z. Are probiotics useful for therapy of Helicobacter pylori diseases? Comp Immunol Microbiol Infect Dis. 2019 Jun;64:99-108. doi: 10.1016/j.cimid.2019.02.010. Epub 2019 Mar 5. PMID 31174707
- [Result] Emara MH, Mohamed SY, Abdel-Aziz HR. Lactobacillus reuteri in management of Helicobacter pylori infection in dyspeptic patients: a double-blind placebo-controlled randomized clinical trial. Therap Adv Gastroenterol. 2014 Jan;7(1):4-13. doi: 10.1177/1756283X13503514. PMID 24381643
- [Result] Yang C, Liang L, Lv P, Liu L, Wang S, Wang Z, Chen Y. Effects of non-viable Lactobacillus reuteri combining with 14-day standard triple therapy on Helicobacter pylori eradication: A randomized double-blind placebo-controlled trial. Helicobacter. 2021 Dec;26(6):e12856. doi: 10.1111/hel.12856. Epub 2021 Oct 10. PMID 34628695